CLINICAL TRIAL: NCT02725307
Title: Non-invasive Peri- and Postoperative Monitoring of Femoral Artery Balloon Angioplasty
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University of Technology (Other); Tampere University (Other)
Responsible Party: Principal Investigator, Niku Oksala, Associate Professor (Tenure track), Tampere University Hospital
Other Study IDs: R15107
Record Dates: First submitted 2016-03-16; First posted 2016-03-31 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Noninvasive pulse wave analysis sensor, ECG-sensor — Noninvasive pulse wave sensors and ECG-sensors are attached

SUMMARY:
This study evaluates a novel noninvasive method to dynamically monitor the effect of percutaneous transluminal angioplasty on arterial pulse wave

DETAILED DESCRIPTION:
Patients with stenosis of superficial femoral artery referred for percutaneous transluminal angioplasty are monitored before, during and after the procedure and pulse wave analysis is conducted.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has been clinically examined at policlinic of vascular surgery
2. The patient has undergone measurement of ankle-brachial index (ABI) and toe-brachial index (TBI) at policlinic of vascular surgery and exhibits abnormal ABI<0.9 or ABI>1.3
3. The patient is considered to have an indication for vascular procedure (critical limb ischemia, intermittent claudication)
4. The patient has been examined with magnetic resonance imaging (MRA)
5. The patient has been considered a candidate for superficial femoral artery percutaneous transluminal balloon angioplasty (PTA) and/or stenting

Exclusion Criteria:

1. Pacemaker
2. Measurement disturbs or risks the subject's treatment process

Withdrawal:

1. Emergency cases
2. By subject's denial
3. Inability to detect signals -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Volunteer patients with diagnosed peripheral atherosclerotic disease referred for femoral artery percutaneous transluminal angioplastu.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-03; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Pulse wave change from baseline during PTA | 1 hour

SECONDARY OUTCOMES:
Pulse wave characteristics after PTA | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Niku Oksala, Assoc. Prof., Principal Investigator — Tampere University
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Undecided